CLINICAL TRIAL: NCT00553241
Title: Phase 1 of Clinical Trial of Risk Factor, Prognosis, Imaging and Standard Management of Transient Ischemic Attack.
Brief Title: Short-Term Prognosis Evaluation of Transient Ischemic Attack Patients Using ABCD2 Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Anzhen Hospital (Other)
Responsible Party: Beijing Anzhen Hospital, Capital Medical University
Other Study IDs: 2007020
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Ischemic Attack, Transient
Keywords: TIA; prognosis; evaluation; management
MeSH Terms: conditions — Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Dept. of Neurology, Beijing Anzhen Hospital, Capital Medical University Beijing 100029, P.R.China
  Every patient admitted to Beijing anzhen hospital with transient ischemic attack will be enrolled in this study, from 06/2007 to 12/2008. duration of the symptom not larger than 1 hour.

SUMMARY:
The purpose of this study is to determine whether the ABCD2 score can be used in patients with transient ischemic attack, admitted to Beijing anzhen hospital, to evaluate the prognosis, risk factor of those patients.

DETAILED DESCRIPTION:
The feasibility of risk stratification of patients with acute transient ischemic attack admitted to Beijing anzhen hospital by the ABCD2 score system is yet to be determined. The aim of this paper was to evaluate and validate the short-term prognosis of TIA patients in Peking area using this new score system.

ELIGIBILITY:
Inclusion Criteria:

* Every patient admitted to Beijing anzhen hospital with transient ischemic attack will be enrolled in this study, from 06/2007 to 12/2008. duration of the symptom not larger than 1 hour.
* Magnetic resonance imaging negative on DWI(no fresh infarction).
* Old infarction or not the criminal infarction.

Exclusion Criteria:

* Patients with hemorrhage stroke were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with transient will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2007-06; Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
end points are defined as follow: transient ischemic attack, stroke, angina, myocardial infraction, peripheral vascular disease, intracerebral hemorrhage and other vascular death. | two year

CONTACTS AND LOCATIONS:
Overall Officials: Qi Bi, Study Chair — Dept. of Neurology, Beijing Anzhen Hospital, Capital Medical University
Locations (1):
- Dept. of Neurology, Beijing Anzhen Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Prabhakaran S, Chong JY, Sacco RL. Impact of abnormal diffusion-weighted imaging results on short-term outcome following transient ischemic attack. Arch Neurol. 2007 Aug;64(8):1105-9. doi: 10.1001/archneur.64.8.1105. PMID 17698700
- [Background] Johnston SC, Gress DR, Browner WS, Sidney S. Short-term prognosis after emergency department diagnosis of TIA. JAMA. 2000 Dec 13;284(22):2901-6. doi: 10.1001/jama.284.22.2901. PMID 11147987
- [Background] Weisberg LA. Clinical characteristics of transient ischemic attacks in black patients. Neurology. 1991 Sep;41(9):1410-4. doi: 10.1212/wnl.41.9.1410. PMID 1891090
- [Background] Albers GW, Caplan LR, Easton JD, Fayad PB, Mohr JP, Saver JL, Sherman DG; TIA Working Group. Transient ischemic attack--proposal for a new definition. N Engl J Med. 2002 Nov 21;347(21):1713-6. doi: 10.1056/NEJMsb020987. No abstract available. PMID 12444191
- [Background] Coull AJ, Lovett JK, Rothwell PM; Oxford Vascular Study. Population based study of early risk of stroke after transient ischaemic attack or minor stroke: implications for public education and organisation of services. BMJ. 2004 Feb 7;328(7435):326. doi: 10.1136/bmj.37991.635266.44. Epub 2004 Jan 26. PMID 14744823
- [Background] Correia M, Silva MR, Magalhaes R, Guimaraes L, Silva MC. Transient ischemic attacks in rural and urban northern Portugal: incidence and short-term prognosis. Stroke. 2006 Jan;37(1):50-5. doi: 10.1161/01.STR.0000195209.26543.8f. Epub 2005 Dec 1. PMID 16322498
- [Background] Clark TG, Murphy MF, Rothwell PM. Long term risks of stroke, myocardial infarction, and vascular death in "low risk" patients with a non-recent transient ischaemic attack. J Neurol Neurosurg Psychiatry. 2003 May;74(5):577-80. doi: 10.1136/jnnp.74.5.577. PMID 12700296
- [Background] Giles MF, Flossman E, Rothwell PM. Patient behavior immediately after transient ischemic attack according to clinical characteristics, perception of the event, and predicted risk of stroke. Stroke. 2006 May;37(5):1254-60. doi: 10.1161/01.STR.0000217388.57851.62. Epub 2006 Mar 30. PMID 16574923
- [Background] Sylaja PN, Coutts SB, Subramaniam S, Hill MD, Eliasziw M, Demchuk AM; VISION Study Group. Acute ischemic lesions of varying ages predict risk of ischemic events in stroke/TIA patients. Neurology. 2007 Feb 6;68(6):415-9. doi: 10.1212/01.wnl.0000252938.76188.52. PMID 17283315
- [Result] Johnston SC, Rothwell PM, Nguyen-Huynh MN, Giles MF, Elkins JS, Bernstein AL, Sidney S. Validation and refinement of scores to predict very early stroke risk after transient ischaemic attack. Lancet. 2007 Jan 27;369(9558):283-92. doi: 10.1016/S0140-6736(07)60150-0. PMID 17258668
- [Result] Tsivgoulis G, Spengos K, Manta P, Karandreas N, Zambelis T, Zakopoulos N, Vassilopoulos D. Validation of the ABCD score in identifying individuals at high early risk of stroke after a transient ischemic attack: a hospital-based case series study. Stroke. 2006 Dec;37(12):2892-7. doi: 10.1161/01.STR.0000249007.12256.4a. Epub 2006 Oct 19. PMID 17053179
- [Result] Rothwell PM, Giles MF, Flossmann E, Lovelock CE, Redgrave JN, Warlow CP, Mehta Z. A simple score (ABCD) to identify individuals at high early risk of stroke after transient ischaemic attack. Lancet. 2005 Jul 2-8;366(9479):29-36. doi: 10.1016/S0140-6736(05)66702-5. PMID 15993230
- [Result] Bray JE, Coughlan K, Bladin C. Can the ABCD Score be dichotomised to identify high-risk patients with transient ischaemic attack in the emergency department? Emerg Med J. 2007 Feb;24(2):92-5. doi: 10.1136/emj.2006.041624. PMID 17251611
- See also: Related Info — http://www.ccmu.edu.cn/english/